CLINICAL TRIAL: NCT00774592
Title: Adolescent Risk Reduction in the Bahamas-Peers and Parents
Brief Title: HIV Risk Reduction in Youth in the Bahamas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bonita Stanton, Professor of Pediatrics, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH069229 (NIH); R01MH069229 (NIH); DAHBR 9A-ASPC (Registry Identifier: Division of AIDS and Health and Behavior Research)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: HIV Infections
Keywords: Adolescent Risk Reduction; HIV/AIDS Prevention; Behavioral Change; HIV
MeSH Terms: conditions — HIV Infections | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental): Focus on Youth in the Caribbean (FOYC) plus Caribbean Informed Parents and Children Together (CImPACT)
  Interventions: Behavioral: FOYC; Behavioral: Caribbean Informed Parents and Children Together (CImPACT)
- 2 (Experimental): FOYC plus Goal For It (GFI)
  Interventions: Behavioral: FOYC; Behavioral: Goal for it (GFI)
- 3 (Active Comparator): Wonderous Wetlands plus GFI
  Interventions: Behavioral: Wonderous Wetlands; Behavioral: Health and Family Life Curriculum (HFLE)
- Grade 10-BFOOY+CImPACT (Experimental): Youth receives HIV intervention; parents receive parental monitoring intervention
  Interventions: Behavioral: Bahamian Focus on Older Youth (BFOOY)
- Grade 10 BFOOY+GFI (Experimental): Youth receive HIV prevention intervention and parents receive attention control intervention on career planning
  Interventions: Behavioral: Bahamian Focus on Older Youth (BFOOY)
- BFOOYand no parent intervention (Experimental): Youth receive HIV prevention intervention; parents receive no intervention
  Interventions: Behavioral: Bahamian Focus on Older Youth (BFOOY)
- Health and FAmily life (Placebo Comparator): Youth receive standard of care (current curriculum); parents receive no intervention
  Interventions: Behavioral: Health and Family Life Curriculum (HFLE)

INTERVENTIONS:
Behavioral: FOYC — FOYC is a face-to-face, eight-session, group behavioral intervention based on protection motivation theory and emphasizing skills and decision-making.
  Arms: 1; 2
Behavioral: Goal for it (GFI) — GFI is a one-session parent intervention consisting of a 20-minute video followed by a discussion regarding the process of setting and reaching goals.
  Arms: 2
Behavioral: Wonderous Wetlands — Wonderous Wetlands is an eight-session, group intervention for youth. It includes field projects and discussions based on ways to save our environment.
  Arms: 3
Behavioral: Caribbean Informed Parents and Children Together (CImPACT) — CImPACT is a parent intervention addressing parental monitoring and communication with youth. It consists of a 20-minute video, a condom practice, and role play simulating a parent-child discussion.
  Arms: 1
Behavioral: Bahamian Focus on Older Youth (BFOOY) — 10 session HIV prevention program
  Arms: BFOOYand no parent intervention; Grade 10 BFOOY+GFI; Grade 10-BFOOY+CImPACT
Behavioral: Health and Family Life Curriculum (HFLE) — Standard Grade 10 curriculum
  Other Names: Standard grade 10 health curriculum
  Arms: 3; Health and FAmily life

SUMMARY:
This study will examine whether pairing a grade 6 in-school HIV education program and a parent training program will reduce prevalence of behaviors that present high risk of HIV infection in youth in the Bahamas.

In a continuation of this study, we shall examine whether an in-school HIV prevention program delivered to grade 10 students reduces HIV risk behavior and the impact of both the grade 6 intervention and the grade 10 intervention compared to the grade 6 intervention alone.

DETAILED DESCRIPTION:
HIV infection in the Bahamas is the leading cause of death among Bahamians between the ages of 15 and 44. It is estimated that 4.13% of adults in the Bahamas are HIV infected, and the Bahamas has the highest annual incidence of AIDS in the English-speaking Caribbean. One cause for these high rates of infection is the prevalence of risky behaviors among Bahamian youth. Among youth between the ages of 13 and 15, 32% are sexually experienced, with that rate rising to 57% among youth age 16 or older. Approximately half of these adolescents have never used birth control, and only one third use birth control consistently.

This study will examine the benefits of combining a youth HIV prevention education program with a parental program focused on communication and monitoring. The youth education program, developed in the United States but modified to address Caribbean culture, is called Focus on Youth in the Caribbean (FOYC). FOYC has already been shown to be effective in increasing condom use, knowledge of HIV, and knowledge of risks associated with unprotected sex and drug use. Including parents in this intervention effort may broaden and sustain its effects. A study of seventh to eleventh graders found that teens were six times less likely to engage in sexual activity if they thought their mothers disapproved of it. The study also found that teens often did not have a clear idea of what their parents approved of or disapproved of, indicating a need for better communication between parents and children. Other studies have shown that parents who monitor their children reduce the likelihood that those children have unprotected sex or use drugs. The parental intervention program, called Caribbean Informed Parents and Children Together (CImPACT), has been shown to increase communication between parents and children and, when paired with a face-to-face intervention, enhance condom skills and lower rates of sex, unprotected sex, cigarette use, and alcohol use. This study will examine whether pairing the FOYC and CImPACT interventions will reduce prevalence of behaviors that present high risk of HIV infection in youth in the Bahamas.

Parents will be randomly assigned to receive either the CImPACT program or a control program called Goal for It (GFI), both of which will be implemented in a 1.5-hour training session. Schools will be randomly assigned to receive either the FOYC program or a control program entitled Wonderous Wetlands. Both programs will be implemented as part of the curriculum in 15 Bahamian elementary schools. Children, therefore, will be part of 1 of 3 groups:

1. Parent receiving the CImPACT program; school receiving the FOYC program
2. Parent receiving the GFI program; school receiving the FOYC program
3. Parent receiving the GFI program; school receiving the Wonderous Wetlands program

Parents and children will be assessed at the beginning of the study and after 6, 12, 18, 24, and 36 months. These assessments will include questionnaires measuring high-risk behaviors, conceptions of risks and rewards involved in high-risk behaviors, and parent and adolescent communication and monitoring.

In the continuation of this study we will:

1. Recruit 2600 youth (and their parents) from 172 Grade 10 FHLE classrooms over two years in all seven government high schools in New Providence, The Bahamas
2. Randomly assign at the level of the classroom 2400 youth (and their parents) from 160 classes to one of four intervention conditions: 1) HFLE only (no parent intervention); 2) BFOOY only (no parent intervention); 3) BFOOY plus ImPACT (delivered to parent-youth dyads); or 4) BFOOY plus GFI (delivered to parent-youth dyads);
3. Randomly assign one of the seven high schools (with ~12 HFLE classes and ~200 students) to a "control school" condition to permit exploration of possible class-to-class contamination within schools
4. Assess intervention effects on the entire youth sample at 6, 12, 18 and 24 months post-intervention and among parents at 6 and 12 months
5. Conduct sub-group analyses to explore: i) the impact of related and intensive interventions received at two critical junctures during adolescence; ii) the effect of being part of a longitudinal trial on risk/protective behaviors; and iii) the extent of intervention contamination when randomization is conducted at the level of the class rather than the school. Subgroups will include: Exposed youth (youth who received FOYC in Grade 6) and Naïve youth (youth who did not receive FOYC in Grade 6); Enrolled youth (youth who were enrolled in the ongoing evaluation of FOYC whether as controls or intervention (FOYC) youth) and Not-enrolled youth (youth who were never part of the ongoing study); and Control School youth (those randomly assigned to the control condition at the level of the school in Year 2) and Control Class youth (those assigned to the control condition at the level of the class)

Intervention effect (primary hypotheses):

1. Youth randomized to HFLE only will exhibit significantly higher rates of HIV risk behavior, intentions and perceptions and lower knowledge and condom skills through 24 months post-intervention than each of the other three groups;
2. Youth randomized to BFOOY plus GFI will exhibit higher rates of abstinence behavior, intentions and perceptions than youth randomized to BFOOY alone through 24 months follow-up
3. Youth randomized to BFOOY plus ImPACT will exhibit lower rates of HIV risk behavior, intentions and perceptions and higher rates of knowledge, condom skills, and STD testing than each of the other three groups through 24 months follow-up; Parents receiving ImPACT will exhibit higher knowledge and condom use skills than GFI or control parents; ImPACT parents and youth will report higher rates of discussion about HIV prevention and safe sex than parents and youth in the other three intervention groups
4. Intervention behavioral effects will be consistent with changes in perceptions and intentions as posited by the PMT, the theoretic model of behavioral change on which BFOOY is based

Secondary/exploratory hypotheses will include:

1. At baseline, Exposed Youth will demonstrate higher rates of condom-use and condom-use intentions and perceptions than Naive youth
2. Exposed youth will demonstrate higher protective behaviors, intentions and perceptions compared to Naive Youth within an intervention category (BFOOY or HFLE) throughout the follow-up period
3. Enrolled youth who received FOYC in Grade 6 will not differ from Not-enrolled youth who received FOYC in Grade 6 with respect to intentions, perceptions and knowledge
4. Youth in the Control Classes will not differ from youth in the Control school with respect to HIV knowledge, perceptions and intentions As a result of this study we shall be able to identify of one or more interventions or intervention combinations targeting mid-adolescents to reduce HIV risk behavior and address questions regarding possible interactions between intervention receipt in both the pre-adolescent and mid-adolescent years. With this knowledge, health policy officials globally, including those in The Bahamas, will be able to make evidence-based decisions appropriate to their resources and the epidemiology of the epidemic in their settings.

ELIGIBILITY:
Inclusion Criteria:

* Attends 1 of the 15 participating Bahamian elementary schools
* Enrolled in grade 6
* Participation of at least 1 parent

In second study:

* Attends 1 of 8 participating government highschools
* Enrolled in grade 10

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction of high-risk behaviors | Measured at baseline and after 6, 12, 18, 24, and 36 months

SECONDARY OUTCOMES:
Intentions concerning high-risk behaviors | Measured at baseline and after 6, 12, 18, 24, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bonita F. Stanton, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University School of Medicine, Detroit, Michigan, United States

REFERENCES:
- [Background] Yu S, Deveaux L, Lunn S, Liu H, Brathwaite N, Li X, Cottrell L, Marshall S, Stanton B. At greatest risk: pre- and early adolescent Bahamian youth experiencing anal intercourse. Int J STD AIDS. 2007 Jun;18(6):396-401. doi: 10.1258/095646207781024784. PMID 17609029
- [Background] Yu S, Marshall S, Cottrell L, Li X, Liu H, Deveaux L, Harris C, Brathwaite N, Lunn S, Stanton B. Longitudinal predictability of sexual perceptions on subsequent behavioural intentions among Bahamian preadolescents. Sex Health. 2008 Mar;5(1):31-9. doi: 10.1071/sh07040. PMID 18361852
- [Background] Gong J, Stanton B, Lunn S, Deveaux L, Li X, Marshall S, Brathwaite NV, Cottrell L, Harris C, Chen X. Effects through 24 months of an HIV/AIDS prevention intervention program based on protection motivation theory among preadolescents in the Bahamas. Pediatrics. 2009 May;123(5):e917-28. doi: 10.1542/peds.2008-2363. Epub 2009 Apr 20. PMID 19380429
- [Background] Chen X, Lunn S, Deveaux L, Li X, Brathwaite N, Cottrell L, Stanton B. A cluster randomized controlled trial of an adolescent HIV prevention program among Bahamian youth: effect at 12 months post-intervention. AIDS Behav. 2009 Jun;13(3):499-508. doi: 10.1007/s10461-008-9511-0. Epub 2008 Dec 31. PMID 19116781
- [Background] Liu H, Yu S, Cottrell L, Lunn S, Deveaux L, Brathwaite NV, Marshall S, Li X, Stanton B. Personal values and involvement in problem behaviors among Bahamian early adolescents: a cross-sectional study. BMC Public Health. 2007 Jul 2;7:135. doi: 10.1186/1471-2458-7-135. PMID 17605792
- [Result] Deveaux L, Stanton B, Lunn S, Cottrell L, Yu S, Brathwaite N, Li X, Liu H, Marshall S, Harris C. Reduction in human immunodeficiency virus risk among youth in developing countries. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1130-9. doi: 10.1001/archpedi.161.12.1130. PMID 18056557
- [Result] Deveaux L, Lunn S, Bain RM, Gomez P, Kelly T, Brathwaite N, Russell-Rolle G, Li X, Stanton B. Focus on youth in the Caribbean: beyond the numbers. J Int Assoc Physicians AIDS Care (Chic). 2011 Sep-Oct;10(5):316-25. doi: 10.1177/1545109710397367. Epub 2011 Mar 23. PMID 21430238
- [Result] Chen X, Stanton B, Gomez P, Lunn S, Deveaux L, Brathwaite N, Li X, Marshall S, Cottrell L, Harris C. Effects on condom use of an HIV prevention programme 36 months postintervention: a cluster randomized controlled trial among Bahamian youth. Int J STD AIDS. 2010 Sep;21(9):622-30. doi: 10.1258/ijsa.2010.010039. PMID 21097734
- [Result] Chen X, Lunn S, Harris C, Li X, Deveaux L, Marshall S, Cottrell L, Stanton B. Modeling early sexual initiation among young adolescents using quantum and continuous behavior change methods: implications for HIV prevention. Nonlinear Dynamics Psychol Life Sci. 2010 Oct;14(4):491-509. PMID 20887691
- [Result] Stanton B, Deveaux L, Lunn S, Yu S, Brathwaite N, Li X, Cottrell L, Harris C, Clemens R, Marshall S. Condom-use skills checklist: a proxy for assessing condom-use knowledge and skills when direct observation is not possible. J Health Popul Nutr. 2009 Jun;27(3):406-13. doi: 10.3329/jhpn.v27i3.3383. PMID 19507756
- [Result] Stanton B, Chen X, Koci V, Deveaux L, Lunn S, Harris C, Brathwaite N, Gomez P, Li X, Marshall S. Effect of a grade 6 HIV risk reduction intervention four years later among students who were and were not enrolled in the study trial. J Adolesc Health. 2012 Mar;50(3):243-9. doi: 10.1016/j.jadohealth.2011.06.012. Epub 2011 Sep 3. PMID 22325129